CLINICAL TRIAL: NCT05442047
Title: Efficacy and Safety of NNC6019-0001 at Two Dose Levels in Participants With Transthyretin Amyloid Cardiomyopathy (ATTR CM)
Brief Title: A Research Study to Look at How a New Medicine Called NNC6019-0001 Works and How Safe it is for People Who Have Heart Disease Due to Transthyretin (TTR) Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6019-4940; U1111-1271-3861 (Other: World Health Organization (WHO)); 2021-006226-49 (EudraCT Number)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Transthyretin Amyloid Cardiomyopathy (ATTR CM)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NNC6019-0001, Dose 1 (Experimental): Participants will receive dose 1 intravenous (i.v.) infusion of NNC6019-0001 every 4 weeks (Q4W) added to standard of care until week 52.
  Interventions: Drug: NNC6019-0001
- NNC6019-0001, Dose 2 (Experimental): Participants will receive dose 2 i.v. infusion of NNC6019-0001 Q4W added to standard of care until week 52.
  Interventions: Drug: NNC6019-0001
- Placebo (Placebo Comparator): Participants will receive i.v. infusion of placebo (NNC6019-0001) Q4W added to standard of care until week 52.
  Interventions: Drug: Placebo (NNC6019-0001)

INTERVENTIONS:
Drug: NNC6019-0001 — Participants will receive i.v infusionof NNC6019-0001.
  Arms: NNC6019-0001, Dose 1; NNC6019-0001, Dose 2
Drug: Placebo (NNC6019-0001) — Participants will receive i.v. infusion of placebo (NNC6019-0001).
  Arms: Placebo

SUMMARY:
This study is testing a potential new medicine, NNC6019-0001, for people who have a heart disease due to TTR amyloidosis.The study will look at if this medicine can reduce the symptoms of a heart disease due to TTR amyloidosis, such as heart failure. Participants will either get NNC6019-0001 (apotential new medicine) or placebo (a medicine which has no effect on the body). Which treatment participants get is decided by chance. The chance of getting NNC6019-0001 is two times higher than getting placebo. NNC6019-0001 is not yet approved in any country or region in the world. It is a new medicine that doctors cannot prescribe yet. Participants will get an infusion of the study medicine 13 times, once every 4 weeks. The study will last for about 64 weeks after the first dose of medicine. Participants cannot participate in this study if they have a heart disease other than a heart disease due to TTR amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age greater than or equal to (>=) 18 to less than (<) 85 years at the time of signing informed consent.
* Have an established diagnosis of Transthyretin amyloid cardiomyopathy (ATTR CM) with either wild-type transhyretin (TTR) or hereditary transthyretin (TTR) genotype as per local standards.
* Expected to be on stable doses of cardiovascular medical therapy 6 weeks prior to the randomisation visit.
* Known end-diastolic interventricular septal wall thickness greater than or equal to (>=) 12 millimeters (mm).
* Presently classified as New York Heart Association (NYHA) Class II-III.
* N-terminal-pro brain natriuretic peptide (NT-proBNP) concentration greater than or equal to (>=) 650 picograms per milliliter (pg/mL) in sinus cardiac rhythm and greater than (>) 1000 pg/mL in atrial fibrillation at screening.
* Completed greater than or equal to (>=) 150 meters to less than or equal to (<=) 450 meters on the 6-minute walk test (MWT) at screening.
* Estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 25 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) at screening.

Exclusion Criteria:

* Cardiomyopathy not primarily caused by transthyretin amyloid cardiomyopathy transthyretin amyloid cardiomyopathy (ATTR CM), for example, cardiomyopathy due to hypertension, valvular heart disease, or ischemic heart disease.
* A prior solid organ transplant.
* Planned solid organ transplant during the study.
* Presence or history of malignant neoplasm (other than basal or squamous cell skin cancer, insitu carcinomas of the cervix, or in-situ/high grade prostatic intraepithelial neoplasia (PIN) or low-grade prostate cancer) within 5 years before screening.
* Current treatment with calcium channel blockers with conduction system effects (example [e.g.], verapamil, diltiazem). The use of dihydropyridine calcium channel blockers is allowed. The use of digoxin will only be allowed if required for management of atrial fibrillation with rapid ventricular response.
* Acute coronary syndrome, unstable angina, stroke, transient ischemic attack (TIA), coronary revascularization, cardiac valve repair, or major surgery within 3 months of screening.
* Body weight >120 kilogram (kg) (264.6 pounds [lb]) at screening.
* History of contrast allergy or adverse reactions to gadolinium-containing agents.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walk test (6-MWT) | From baseline (week 0) to visit 15 (week 52)
  Measured in Meters
Change in N-terminal-pro brain natriuretic peptide (NT-proBNP) | From baseline (week 0) to visit 15 (week 52)
  Measured in Percentage

SECONDARY OUTCOMES:
Change in myocardial extracellular volume (ECV) | From baseline (week 0) to visit 15 (week 52)
  Measured in Percentage (%)-points
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score (CSS) | From baseline (week 0) to visit 15 (week 52)
  The KCCQ is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and health-related quality of life limitation from heart failure. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. CSS scores range from 0 to 100 and lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Change in neuropathy impairment score (NIS) | From baseline (week 0) to visit 15 (week 52)
  NIS is a clinical assessment that tests muscle strength, reflex activity, and sensation of toes and fingers, and can be used to assess neurologic function in hereditary transthyretin amyloid (hATTR). The total NIS score is graded on a scale of 0-244, with a higher score indicating greater impairment.
Change in troponin I | From baseline (week 0) to visit 15 (week 52)
  Measured in nanogram per milliliter (ng/mL)
Change in global longitudinal strain (GLS) on echocardiography | From baseline (week 0) to visit 15 (week 52)
  Measured in Percentage (%)-points
Number of treatment emergent adverse events | From baseline (week 0) to visit 16 (week 64)
  Measured as Events
Time to occurrence of all-cause mortality | From baseline (week 0) to visit 16 (week 64)
  Measured in Weeks
Number of cardiovascular (CV) events comprising hospitalisation due to CV events or urgent heart failure visits | From baseline (week 0) to visit 16 (week 64)
  Measured as Events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency 2834, Study Director — Novo Nordisk A/S
Locations (35):
- United States (9):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Cedars-Sinai Medical Center_Los Angeles, Beverly Hills, California
  - Stanford Hlth Cre-Boswell Clin, Stanford, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - NW Univ-Bluhm Cardiovasc Inst, Evanston, Illinois
  - Univ of MD Schl of Med, Baltimore, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Oregon Hlth Sci Univ-Portland, Portland, Oregon
- Canada (2):
  - University of Calgary_Cardiology, Calgary, Alberta
  - Ctr for Cardiovascular Innovation, Vancouver, British Columbia
- II. interni klinika VFN - Kardiologie a angiologie, Prague, Czechia
- France (3):
  - Ap-Hp-Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-1, Toulouse
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-1, Toulouse Cedex 9 TSA 50032
- Germany (5):
  - UniklinikHeidelberg - Innere Med. III - Kardiologie, Angiologie, Pneumologie, Heidelberg
  - LMU Klinikum München Klinik und Poliklinik 1, München
  - Universitätsklinikum Münster - Klinik für Kardiologie I, Münster
  - Universitatsklinikum Wurzburg AöR, Würzburg
  - Universitatsklinikum Würzburg - Zentrum für Herzinsuffizienz, Würzburg
- Italy (2):
  - Fondazione Toscana Gabriele Monasterio - Dipartimento Cardiotoracico - UOC Cardiologia e Medicina Cardiovascolare, Pisa, Pi
  - Centro per lo Studio e la Cura delle Amiloidosi Sistemiche Fondazione IRCCS Policlinico San Matteo, Pavia, PV
- Japan (6):
  - Hospital of the University of Occupational and Environmental Health, Cardiology, Nephrology, Fukuoka
  - Hiroshima University hospital, Cardiovascular Medicine, Hiroshima
  - Kumamoto University Hospital, Cardiovascular Medicine, Kumamoto-shi, Kumamoto
  - Shinshu University Hospital, Department of Neurology, Nagano
  - Nagasaki University Hospital, Cardiovascular Medicine, Nagasaki
  - Okayama University Hospital_Cardiovascular Medicine, Okayama-shi, Okayama
- Netherlands (2):
  - UMC Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Portugal (3):
  - Hospital da Senhora da Oliveira - Guimarães, Guimarães
  - Unidade Local de Saude do Alto Ave, E.P.E., Guimarães
  - Unidade Local De Saude De Tras-Os-Montes E Alto Douro E.P.E., Vila Real
- Spain (2):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Fontana M, Garcia-Pavia P, Grogan M, Shah SJ, Engelmann MDM, Hovingh GK, Kristen AV, Lim-Watson MZ, Malling B, Kar S, Revanna M, Sarswat N, Tsujita K, Alexander KM, Maurer MS. Coramitug, a Humanized Monoclonal Antibody for the Treatment of Transthyretin Amyloid Cardiomyopathy: A Phase 2, Randomized, Multicenter, Double-Blind, Placebo-Controlled Trial. Circulation. 2026 Jan 27;153(4):214-225. doi: 10.1161/CIRCULATIONAHA.125.077304. Epub 2025 Nov 10. PMID 41212997
- [Derived] Suhr OB, Grogan M, Silva AMD, Karam C, Garcia-Pavia P, Drachman B, Zago W, Tripuraneni R, Kinney GG. PRX004 in variant amyloid transthyretin (ATTRv) amyloidosis: results of a phase 1, open-label, dose-escalation study. Amyloid. 2025 Mar;32(1):14-21. doi: 10.1080/13506129.2024.2420809. Epub 2024 Oct 29. PMID 39472768